CLINICAL TRIAL: NCT04643951
Title: Pain in Pediatric Dentistry - a Grounded Theory Study on the Experiences of Dental
Brief Title: Pain in Pediatric Dentistry - a Grounded Theory Study on the Experiences of Dental Professionals and Students
Status: Recruiting | Type: Observational
Sponsor: Malmö University (Other)
Responsible Party: Principal Investigator, Rikard Roxner, Principal investigator, Malmö University
Other Study IDs: FO 2020/529.
Record Dates: First submitted 2020-11-09; First posted 2020-11-25 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Dental students: Dental students in their two final years. No intervention.
  Interventions: Behavioral: Interview
- Dental professionals: Dental professionals aged 18-65, regularly working with children. No intervention.
  Interventions: Behavioral: Interview

INTERVENTIONS:
Behavioral: Interview — Interview study using Grounded theory, to investigate dental professionals' and students' perception of child patient's experience and need for treatment regarding procedural and postoperative pain.

SUMMARY:
This is a qualitative interview study, using Grounded Theory. The aim is to deepen our knowledge about how the dental team (dentists, dental hygienists, and dental assistants) and dental students perceive child patients' pain and how they perceive they are equipped to prevent and deal with child patients' pain and the child's response to pain during and after dental treatment.

DETAILED DESCRIPTION:
BACKGROUND Pain in conjunction with dental treatment should be avoided, especially when treating children. Many dental procedures may result in procedural and/or postoperative pain. There is a well-documented relationship between perceived pain during dental treatment, and the development of dental fear and anxiety. This may lead to suffering for the patient, avoidance of dental care, and increasing treatment costs for the individual and society. Dental care professionals are responsible for providing as painless dental treatments as possible to their child patients. Earlier studies have pointed towards an underusage of local anesthetics when providing dental care to children. Though previous studies have not been able to fully answer why this is. Thus, the aim of this study is to gain knowledge into how dental professionals and students experience and relate to the child patient's experience of pain during and after dental treatment.

METHOD This is a qualitative study using Grounded Theory (GT). Dental students in their last two years of education and dental professionals (dentists, dental hygienists, and dental assistants), will be consecutively enrolled after signing an informed consent form.

In-depth interviews of approximately one hour each will be performed with the informants at a place of their convenience. Appropriate measures will be taken regarding public health recommendations in effect due to the Covid-19 pandemic.

In GT no sample size calculation is done. Participants will be included until saturation in data is reached, i.e. no new information can be obtained from further interviews. In GT this is often achieved after 10-15 interviews, but due to the scope of this study involving several different professionals and students it is likely the number of informants will be closer to 25. All interviews will be tape recorded, and without delay, the interviews will be transcribed verbatim. Data analyses and data collection will be done in tandem. The transcribed interviews will be analyzed, and codes identified. These codes will then be merged into different preliminary categories. In the following axial coding process, each category will be further developed by identifying common dimensions and characteristics (subcategories). Relations between data and categories is sought, and hereby a new whole is created. Selective coding will lead to data saturation and validation. Saturation can also be achieved by already retrieved data being re-coded.

KNOWLEDGE GAINS GT is a theory generating method. This is especially suitable for research areas where theories are scarce or lacking. A lot of research within the medical and dental field today, takes the perspective of the investigator, and far too seldom is the subjective experience of those directly affected (e.g. professionals and/or patients) heard. From this study we will gain new knowledge into dental professionals' and students' perception of the child patients' experiences of procedural and postoperative pain. These knowledge gains will be important for future research strategies related to pain. In the longer run the results can help lead to a better training of undergraduate students and professionals.

CHANGES TO ORIGINAL STUDY PLAN After the initial interviews were made, we saw that dental students had a pedagogical focus in their interviews. Therefore, we decided to split informants into two groups - dental students and dental professionals. Findings will be presented in two separate scientific papers, one for each group of participants. Interviews with dental students have been completed, while interviews with dental professionals are ongoing.

ELIGIBILITY:
Inclusion Criteria:

* Dental students in their 4th or 5th year of training
* Dental professionals working with child patients on a regular basis

Exclusion Criteria:

• Do not understand Swedish language

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 4th and 5th year dental students, and dental professionals (dentists, dental hygienists, dental assistants)
Sampling Method: Non-Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Pain in pediatric dentistry, a Grounded theory study on the experiences of dental professionals and students. | June, 2021
  By means of in-depth interviews and data analysis according to Grounded Theory, investigate dental professionals' and dental students' perceptions of child patients' experiences of pain related to dental treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Gunilla Klingberg, Prof., Study Chair — Malmö University
Locations (1):
- Malmö University, Malmo, Skåne County, Sweden

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Berlin H, List T, Ridell K, Klingberg G. Dentists' attitudes towards acute pharmacological pain management in children and adolescents. Int J Paediatr Dent. 2018 Mar;28(2):152-160. doi: 10.1111/ipd.12316. Epub 2017 Jul 10. PMID 28691744
- [Background] Murtomaa H, Milgrom P, Weinstein P, Vuopio T. Dentists' perceptions and management of pain experienced by children during treatment: a survey of groups of dentists in the USA and Finland. Int J Paediatr Dent. 1996 Mar;6(1):25-30. doi: 10.1111/j.1365-263x.1996.tb00204.x. PMID 8695586
- [Background] Rasmussen JK, Frederiksen JA, Hallonsten AL, Poulsen S. Danish dentists' knowledge, attitudes and management of procedural dental pain in children: association with demographic characteristics, structural factors, perceived stress during the administration of local analgesia and their tolerance towards pain. Int J Paediatr Dent. 2005 May;15(3):159-68. doi: 10.1111/j.1365-263X.2005.00635.x. PMID 15854111
- [Background] Charmaz, K. Grounded theory. In: Smith, J.A., Harre, R. & van Langenhove, L. (eds.) Rethinking methods in psychology. 2nd ed. London: Sage Publications, 1995; 27-49.
- [Background] Glaser, B. & Strauss, A. The discovery of grounded theory: strategies for qualitative research. New York: Aldine de Gruyter, 1967.